CLINICAL TRIAL: NCT01656057
Title: The Impact of Gall Bladder Emptying and Bile Acids on the Human GLP-1-secretion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Filip Krag Knop (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Filip Krag Knop, MD, Ph.D., University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: GALINKUR
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: To Assess the Impact of Bile Acids on Human Glukagon-like-peptide-1 Secretion
Keywords: Bile acids; Gall bladder emptying; Human; Glucagon like peptide 1; GLP-1
MeSH Terms: interventions — Acetaminophen; Metformin; Colesevelam Hydrochloride; desulfated sincalide; Sincalide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Acetaminophen+saline (Experimental): Acetaminophen tablet 1500 mg via nasogastric tube + i.v. saline
  Interventions: Drug: Acetaminophen; Other: Saline
- Acetaminophen+CCK (Experimental): Acetaminophen tablet 1500 mg via nasogastric tube + iv. CCK-8, 24 pmol/kg/hour
  Interventions: Drug: Acetaminophen; Other: Cholecystokinin-8
- Metformin+saline (Experimental): Metformin tablet 1500 mg + Acetaminophen tablet 1500 mg via nasogastric tube + i.v. saline
  Interventions: Drug: Acetaminophen; Drug: Metformin; Other: Saline
- Metformin+CCK (Experimental): Metformin tablet 1500 mg + Acetaminophen tablet 1500 mg via nasogastric tube + iv. CCK-8, 24 pmol/kg/hour
  Interventions: Drug: Acetaminophen; Drug: Metformin; Other: Cholecystokinin-8
- Colesevelam+saline (Experimental): Colesevelam tablet 3750 mg + Acetaminophen tablet 1500 mg via nasogastric tube + iv. saline
  Interventions: Drug: Acetaminophen; Drug: Colesevelam; Other: Saline
- Colesevelam+CCK (Experimental): Colesevelam tablet 3750 mg + Acetaminophen tablet 1500 mg via nasogastric tube + iv. CCK-8, 24 pmol/kg/hour
  Interventions: Drug: Acetaminophen; Drug: Colesevelam; Other: Cholecystokinin-8

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen dissolved in 50 ml of water
  Other Names: Paracetamol
Drug: Metformin — Metformin + acetaminophen dissolved in 50 ml of water
  Arms: Metformin+CCK; Metformin+saline
Drug: Colesevelam — Colesevelam + acetaminophen dissolved in 50 ml of water
  Arms: Colesevelam+CCK; Colesevelam+saline
Other: Cholecystokinin-8 — iv. infusion of CCK-8, 24 pmol/kg/hour for the first 60 minutes
  Other Names: CCK-8
  Arms: Acetaminophen+CCK; Colesevelam+CCK; Metformin+CCK
Other: Saline — iv. saline infusion 40 ml/hour for the first 60 minutes
  Arms: Acetaminophen+saline; Colesevelam+saline; Metformin+saline

SUMMARY:
The last couple of years it has been shown that bile acids not only acts as simple emulsifiers of fat, but constitutes a complex metabolic integrator which not only have an influence on fat digestion and lipid metabolism, but also modulates the energy expenditure in (brown) adipose tissue and muscle tissue. This action is due to stimulation of the receptor TGR5 by bile acids. Recently scientists have discovered that this receptor in rodents is also expressed on the surface of intestinal L-cells (which normally secrets Glucagon-Like Peptide-1 (GLP-1) in response to nutrient stimulation). The stimulation of this receptor has shown a GLP-1 secretion from the intestinal cells which is interesting since GLP-1 has a central role in maintaining normal glucose tolerance and thus blood sugar. Given the above, bile acids has an important impact on intestinal GLP-1 secretion. Whether these scientific findings can be proven in human beings is uncertain.

The primary hypothesis is that stimulating gall bladder emptying via Cholecystokinin (CCK) in healthy subjects will result in a significant GLP-1 response. We also hypothesize that adding orally Metformin or a sequestrant ("a bile acid binder") will further enhance this GLP-1 response.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c < 6,0%
* Not anaemic
* Written informed consent

Exclusion Criteria:

* Liver disease
* Nephropathy
* fasting plasma glucose > 5,6mM
* Diabetes running in the family (parents or grandparents)
* Any medical treatment
* A former medical history of liver- or bile disease
* any surgical procedure conducted in the abdomen
* Body mass index < 18,5 kg/m2 or > 25 kg/m2

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
GLP-1 response as incremental area under curve (iAUC) | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240

SECONDARY OUTCOMES:
Insulin | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240

OTHER OUTCOMES:
c-peptide | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240
glucagon | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240
Glucagon-Like Peptide-2 | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240
Peptide YY | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240
Oxyntomodulin | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240
Glucose-Dependent Insulinotropic Peptide | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240
Bile acids | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240
Gastrin | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240
CCK | -30, -15, 0, 10, 20, 30, 40, 50, 60, 90, 120, 150, 180, 240
Gall bladder emptying assessed ultrasonically | -30, -15, 20, 40, 60, 90, 120, 150, 180
Resting energy expenditure | -10, 50, 210
Estimation of satiety via visual analogue scale | 0, 30, 60, 90, 120, 150, 180, 240

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Rohde, MD, Principal Investigator — Diabetic Research Division, Department of Internal Medicine, University Hospital of Copenhagen, Gentofte Hospital
Locations (1):
- University Hospital of Copenhagen, Gentofte Hospital, Diabetic Research Division, Copenhagen, Hellerup, Denmark

REFERENCES:
- [Derived] Rohde U, Sonne DP, Christensen M, Hansen M, Bronden A, Torang S, Rehfeld JF, Holst JJ, Vilsboll T, Knop FK. Cholecystokinin-Induced Gallbladder Emptying and Metformin Elicit Additive Glucagon-Like Peptide-1 Responses. J Clin Endocrinol Metab. 2016 May;101(5):2076-83. doi: 10.1210/jc.2016-1133. Epub 2016 Mar 22. PMID 27003305